## STUDY PROTOCOL

**Official Title:** Effect of Menstrual Cycle on Postoperative Sensitivity and Rebound Pain in Posterior Composite Restorations: A Double-Blind Split-Mouth Clinical Study

Unique Protocol ID: FIRAT-DENTISTRY ADEMGOK-001

**NCT ID:** .....

Date: 01.09.2022

Principal Investigator: Adem GÖK, DDs, PhD, Assistant Professor

**Affiliation:** Firat University, Faculty of Dentistry, Department of Restorative Dentistry,

Elazig, Turkey

**⊆ mail** agok@firat.edu.tr **C Phone:** +905444142458

### **Study Objectives:**

- **Primary Objective:** To evaluate the effect of menstrual cycle phases on postoperative sensitivity (POS) following direct posterior composite restorations.
- **Secondary Objective:** To assess whether menstrual cycle phases influence the incidence or severity of rebound pain (RP) after inferior alveolar nerve block (IANB).

## **Study Design:**

- Type: Double-blind, split-mouth, randomized clinical trial
- Study Groups:
  - Menstrual Phase Group (MPG): Restorations performed during days 1-3 of menstruation.
  - Ovulatory Phase Group (OPG): Restorations performed on days 11-16, depending on cycle length.
- Number of Participants: 35 women, each receiving two restorations
- **Total:** 70 restorations).
- Masking(Blinding):
  - The operator performing the restorations and the researcher assessing the outcomes were blinded to menstrual cycle phases.

## **Eligibility Criteria:**

### **Inclusion Criteria:**

- Women aged 18-45 years
- Regular menstrual cycles (26-32 days)
- No hormonal contraceptive use
- Vital posterior mandibular molar teeth requiring restorative treatment
- Good oral and periodontal health

#### **Exclusion Criteria:**

- Irregular menstrual cycles or hormonal disorders
- Pregnancy or lactation
- Use of analgesics or anti-inflammatory drugs within 48 hours before treatment
- Severe periodontal disease or need for endodontic treatment

#### **Interventions & Procedures:**

- **Anesthesia:** Inferior alveolar nerve block (**IANB**) with articaine hydrochloride with epinephrine (1:100,000)
- **Restorative Material:** Clearfil Universal Bond Quick (Kuraray, Japan) and Clearfil Majesty Posterior (Kuraray, Japan).
- Postoperative Sensitivity (POS) Assessment:
  - o VAS (0-10) measured at Day 1, Day 2, and Day 3 after restoration.
- Rebound Pain (RP) Assessment:
  - o VAS (0-10) measured at Hour 4, Hour 8, and Hour 12 after anesthesia resolution.

# **Statistical Analysis:**

- Cochran's Q test for intragroup comparisons
- McNemar's test for post-hoc analysis
- Chi-Square test or Fisher's Exact Test for intergroup comparisons
- **Bonferroni correction** for multiple comparisons
- Significance Level: p < 0.05

## **Ethical Approval:**

- Non-Interventional Research Ethics Committee of Firat University
- Reference No: 2022/08-07
- ClinicalTrials.gov Registration No: has not been created yet

Date of creation: 01.09.2022